CLINICAL TRIAL: NCT02986945
Title: Community-Partnered Participatory Development of Mobile Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHINO 2013-0834
Record Dates: First submitted 2016-12-01; First posted 2016-12-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Depressive Symptoms
Keywords: Depressive symptoms; resiliency; Health Promotion; minority health; text-messaging app; participatory technology development
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Experimental): Resiliency App: Study participants randomized to the Immediate group will receive the text-messaging app, B-RESILIENT-an adaptation of a Resiliency Course for improving mood in individuals with depressive symptoms--for 4 weeks.
  Wk 1: BOOST - manage unhealthy thoughts. Wk 2: BREAK - doing pleasant activities. Wk 3: BUDDY - effective communication for social support. Wk 4: Review of first 3 weeks. Each day, users will receive a daily affirmation text message, a series of approximately 5-10 text messages on the topic of the day, and a daily goal corresponding to the day's content (e.g. do a pleasant activity). At the end of the day, users will receive text messages asking them to report whether they completed the daily goal, followed by a daily mood measure.
  Interventions: Behavioral: Resiliency App
- Delayed (Other): Resiliency App: The Delayed arm will receive the intervention after the Immediate Arm completes its use of the intervention.
  Interventions: Behavioral: Resiliency App

INTERVENTIONS:
Behavioral: Resiliency App
  Other Names: B-RESILIENT

SUMMARY:
The purpose of the study is to test an experimental method, a text-messaging app called B-RESILIENT, for improving participants' mood. B-RESILIENT is a text messaging app adaptation of a Resiliency Course, developed by community members known as Building Resiliency and Community Hope.

DETAILED DESCRIPTION:
In phase 1, the investigators held a series of in-person and virtual workshops with the Partnered Research Center for Quality Care (PRC) community partners to co-develop mobile interventions to address community priorities. The goal of the workshops was to develop novel mobile interventions based on stakeholder input. The specific intervention to be developed was determined based on stakeholder input regarding community priorities during the workshops. Workshops were audio and/or video recorded to document the process. One of the tools used in this process was the Chorus Participatory Mobile Framework created at the Center for Health Services and Society at UCLA. Chorus is a web application that allows users to easily create mobile (text messaging and interactive voice) applications in real-time without requiring any server programming. The investigators used this framework during the workshops to develop and test the application in real-time. Participants were also given phone numbers to call or text in to the intervention that they co-developed for the purpose of testing, providing feedback, and guiding future development.

In phase 2, the investigators will conduct a pilot randomized control trial of the B-RESILIENT tool developed during the workgroup phase 1. Investigators will enroll 30 adults in South Los Angeles to participate in a randomized, wait-list trial. The study group will receive the intervention for 4 weeks, followed by the wait-list group for another 4 weeks. Investigators will conduct baseline and follow-up surveys, as well as in-person or telephone workgroups, to assess the tool's usability and feasibility for supporting management of mood and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Speak English
3. Endorse one item on the PHQ-2
4. Are able to be contacted by phone or email, and have a cell phone that receives text messages
5. Have internet access

Exclusion Criteria:

1. Under age 18 years
2. Endorse no items on PHQ-2 screener
3. PHQ-8 score of 15 or greater on the baseline interview
4. No cell phone and internet access
5. Currently homeless
6. Has a prior diagnosis of schizophrenia, psychosis, bipolar disorder
7. Current alcohol and substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Depressive symptom count as measured by the Patient Health Questionnaire 8 | Change from baseline at 1 month
  The Patient Health Questionnaire (PHQ) 8 is a standard measure of depressive symptoms.

OTHER OUTCOMES:
Fordyce Emotions Questionnaire | Change from baseline at 1 month
  This questionnaire assesses current happiness with four questions. The first question assesses current happiness on a scale of 0 (extremely unhappy) to 10 (extremely happy). Questions 2 through 4 asks the percent of time the respondent feels happy; percent of time unhappy; and percent of time neutral.
Brief Resilience Scale | Change from baseline at 1 month
  A 6 item measure of the ability to bounce back or recover from stress.
Coping Strategies | Change from baseline at 1 month
  The coping strategies questionnaire is a 4 item measure used to determine any use of avoidant and/or active coping strategies to stressful situations or problems.
Social Supports | Change from baseline at 1 month
  The social support survey is a 10 item measure created to help assess various dimensions of social support (emotional, affectionate, and positive social interaction).
Employment, work missed for those employed | Change from baseline at 1 month
  The employment questionnaire has 1 item that assesses the employment situation of participants. There are 4 additional items reporting any days missed of work.
Income | Change from baseline at 1 month
  The income survey is a 1 item measure created to evaluate the level of income within each household.
Client Use of Services | Change from baseline at 1 month
  The client use of services Scale is an 6 item measure that assesses access to and use of general health services in the community. This includes hospitalizations, ER visits, Mental Health Services, Social and Community-based Services, and other trusted locations.
Current Medication Use | Change from baseline at 1 month
  The current medication use is a measure with 2 items created to identify any prescribed medications being consumed for mental or emotional problems such as depression, anxiety, or nerves.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O'Hora, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Healthy African American Families, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No